CLINICAL TRIAL: NCT05282199
Title: Efficacy of Inspiratory Muscle Training (IMT) on Sleep Quality, Exercise Tolerance and Pulmonary Radioaerosol Deposition Pattern in Post COVID-19 Infection Subjects
Brief Title: Inspiratory Muscle Training in Post COVID-19 Infection Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, José Carlos Nogueira Nóbrega Júnior, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMT and COVID-19
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: COVID-19; Inspiratory muscle training; scintigraphy; radioaerosol distribution; inhalation therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMT group (Experimental): In the group of post-COVID patients in which reduced endurance and inspiratory muscle power are identified, inspiratory muscle training (IMT) will be performed with a load equivalent to 50% of MIP (assessed weekly) for eight weeks.
  Interventions: Other: INSPIRATORY MUSCLE TRAINING

INTERVENTIONS:
Other: INSPIRATORY MUSCLE TRAINING — In the group of post-COVID-19 patients in which reduced endurance and inspiratory muscle power are identified, inspiratory muscle training (IMT) will be performed with a load equivalent to 50% of MIP (assessed weekly) for eight weeks.
  Other Names: Powerbreath® ClassicLight

SUMMARY:
Long-term COVID has been considered a clinical condition in which the patient, after the critical period of the disease, still has systemic symptoms such as muscle weakness, inability to exercise, sleep disorders and it is still unknown what happens to the pulmonary deposition process. of aerosols. In clinical practice, inspiratory muscle training has been used to treat these patients, but the effectiveness of this intervention in reducing these symptoms is still considered a gap in the literature. To evaluate the effectiveness of inspiratory muscle training in individuals who were affected by COVID-19 to improve submaximal aerobic capacity, respiratory muscle strength, sleep quality, pulmonary deposition of the inhaled radiopharmaceutical and quality of life. This is a quasi-experimental study. , in which elderly volunteers over 18 years of both sexes residing in the city of Recife-Pernambuco will participate. The sample will consist of individuals who have been affected by COVID-19, whose severity of the disease will be classified according to the criteria established by the study by Parasher (2020). 6 minutes. The pulmonary deposition of the radiopharmaceutical will be evaluated pulmonary function will be evaluated by scintigraphy while the maximum respiratory pressures will be evaluated by a manovacuometer. Subjective sleep assessment will be assessed using the Pittsburgh Sleep Quality Index (PSQI) and the Epworth Daytime Sleepiness Scale (ESS) and objective measurement by actigraphy. Finally, quality of life will be measured by the generic Medical OutcomesStudy 36-Item Short-Form HealthSurvey (SF-36) questionnaire. In the group of post-COVID patients in which the reduction in endurance and inspiratory muscle power are identified, an inspiratory muscle training (IMT) will be performed with a load equivalent to 50% of the MIP (assessed weekly), for eight weeks.

DETAILED DESCRIPTION:
The pulmonary function test will be used for the inclusion criteria and characterization of the sample. The Medical Microloop spirometer will be used. The test will be performed at least three times, respecting an interval of at least one minute between maneuvers, until the device considers the best maneuver as reproducible and acceptable. Subjects will perform manovacuometry before and weekly until completing 8 weeks of IMT. The present study will follow the recommendations proposed by the ThoracicSociety/ EuropeanRespiratorySociety (ATS/ERS) and the Brazilian Society of Pneumology and Tisiology (SBPC), thus, during the collection of the values referring to MIP, the patient will be seated, with free arms and will be guided by the person responsible for carrying out the test to attach a mouthpiece (divers type) with a leak orifice of 2mm of internal diameter to his mouth, the individual will be instructed to maintain an inspiratory and expiratory pressure for at least 1.5s so that it can be observed the maximum sustained pressure for one second (maximum mean pressure) in the manovacuometer (MVD 300, Globalmed, Brazil), used in the Cardiopulmonary Laboratory of the Department of Physiotherapy of the Federal University of Pernambuco. The measures with the highest value presented will be used (with variation less than or equal to 10% among the others).

The evaluation of measures of inspiratory muscle performance will be performed before and after the 8 weeks of training. The Test of Incremental Respiratory Endurance (TIRE) provides a more comprehensive assessment of inspiratory musculature by measuring not only strength, but also endurance and work capacity in a single session. The TIRE includes measurements of MIP (MIP), Maximum Sustained Inspiratory Pressure (SMIP) and Inspiratory Duration (DI). A single assessment session will consist of 3-5 sequential trials with 60 second rest intervals between efforts. The highest SMIP will be used to identify the best of the repeated attempts within the session, providing the MIP and SMIP values to be documented and used for study purposes. All inspiratory maneuvers will be performed with subjects seated in a chair and using nose clips in accordance with American ThoracicSociety (ATS) standards for respiratory muscle testing. For the objective assessment of objective sleep parameters, actigraphy will be used, which is a method of objective assessment of the sleep-wake cycle and motor activity, based on limb movements for 24 hours. An actigraph (Fitbit) will be placed on the non-dominant wrist (like a wristwatch) to perform movement detection. Data will be collected for 7 consecutive days and, during this period, participants will sleep at home and be asked to adhere to their normal daily activities and sleep-wake schedules. The ESS will be applied before and after the 8 weeks of inspiratory muscle training. It is a scale containing eight daily situations requesting a self-assessment of the individual about the chance of dozing in the execution of these activities, scoring from 0 to 3, where 0: no chance of dozing, 1: small chance, 2: moderate chance, 3: high chance. When the sum of the scale components reaches a value ≥10, it means that the patient has excessive daytime sleepiness that needs to be investigated. The PSQI will be applied before and after the 8 weeks of inspiratory muscle training. It consists of a self-assessment questionnaire, which investigates sleep quality and disturbances over a period of 1 month. It consists of nineteen individual items that give rise to seven scoring "components": subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The SF36 will be applied before and after the 8 weeks of inspiratory muscle training. It consists of a generic instrument for assessing quality of life, which is easy to administer and understand.

The 6MWT will be performed before and after 8 weeks of inspiratory muscle training. Patients will be instructed to walk as quickly as possible in an open and linear corridor of 30m in length, signposted meter by meter. During the walk test, patients will have their SpO2 and HR monitored using a transcutaneous pulse oximeter. The tests will be interrupted if there are symptoms of dyspnea and/or muscle pain, the presence of a suffering face and/or a drop in SpO2 ≤ 88%, with a time counting up to six minutes. It is important to emphasize that pulmonary scintigraphy is a routine examination in the follow-up of patients with ventilation/perfusion disorders.

It is important to emphasize that pulmonary scintigraphy is a routine examination in the follow-up of patients with ventilation/perfusion disorders. Technetium-99m-labeled diethylnotriaminopentaacetic acid (Tc 99m and DTPA) at an activity of 1 millicuri in 0.9% saline for a total volume of 3 ml will be inhaled. For inhalation, an orofacial mask or mouthpiece (Vital signs, West SuSex, UK) fitted with one-way valves and with an inspiratory limb connected to a radioisotope nebulizer (Ventis® II Medical Device, Class II, CE 0459, Ventibox / CIS BioInternational, France) will be used. used.

The inhalation of the radioaerosol will be performed with the individual in a sitting position for the time necessary for the solution to be completed. Subjects will be previously instructed to breathe slowly and deeply through the mouth, performing an inspiratory pause for 3s with each breath. After inhalation, participants will be instructed to rinse their mouths and drink water to clear the throat and esophagus of radioaerosol deposited in these regions. Scintigraphy will be performed before and after the 8 weeks of training. Volunteers will undergo examinations at the Advanced Nuclear Medicine Diagnostic Imaging Clinic with a Nuclear Medicine Specialist. Upon completion of aerosol inhalation, volunteers will be seated in front of the gamma camera (STARCAM 3200 AC/T GE MEDICAL SYSTEMS - UK ) for image acquisition of the posterior thorax for a period of 300 seconds with a matrix of 256 x 256 pixels. After the first image, the collimator will be repositioned to acquire the upper airway/face images. To determine the inhaled mass, the sum of the numbers of counts present in each compartment will be evaluated.

For image analysis, pulmonary and extrapulmonary regions of interest (ROI) will be delimited using the Xeleris 3 Functional Workstation Image software (GE Healthcare, Milwaukee, USA).

Subjects will perform training with moderate load at 50% of MIP. The training will be carried out using the powerbreath®ClassicLight device.

The patient will be instructed to perform the training seated, with knees and ankles flexed at 90º, feet flat on the floor, with one hand holding the device and the other resting on the leg. The nose clip will be placed and the individuals will perform three cycles of 30 respiratory incursions in an explosive way, respecting the one-minute interval between the series. The training will be performed by the patient at home, independently, twice a day, seven days a week, for eight weeks, noting the frequency and any occurrences during the training in the training diary that each individual will receive. The adjustment will be carried out weekly in face-to-face meetings (once a week) in the laboratory and patient monitoring will also be carried out via telephone, through calls made by the responsible researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders, over 18 years of age, who are not undergoing any type of post-infection treatment, with a diagnosis through RT-PCR positive for the Coronavirus, who fall within the period of up to 10 days after hospital discharge will be included. .

Exclusion Criteria:

* Individuals with previous orthopedic, neurological problems or any cardiovascular or respiratory disease in their clinical history, pregnant women and patients in the active phase of infection for the coronavirus, or who cannot maintain proper positioning during the scintigraphy exam will be excluded pulmonary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Radioaerosol Pulmonary Deposition | 3 minutes
  Amount of radiodrug deposited in the lungs after inhalation

CONTACTS AND LOCATIONS:
Overall Officials: ARMELE DORNELAS DE ANDRADE, PhD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not